CLINICAL TRIAL: NCT01038453
Title: Effects of Vitamin D Supplement Before and During Pregnancy on Complications, Birth Weight and Bone Mineral Density During Lactation
Brief Title: Effects of Vitamin D Supplement Before and During Pregnancy on Birth Weight
Acronym: Gravita
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M-20090097
Record Dates: First submitted 2009-12-18; First posted 2009-12-24 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Birth Weight; Vitamin D Deficiency; Pregnancy
MeSH Terms: conditions — Birth Weight; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cholecalciferol (Vitamin D3) 35 µg (Active Comparator): Dietary Supplement: Cholecalciferol (Vitamin D3) 35 µg per day
  Interventions: Dietary Supplement: Cholecalciferol 35 µg per day
- Cholecalciferol (Vitamin D3) 70 µg (Active Comparator): Dietary supplement: Cholecalciferol (Vitamin D3) 70 µg per day
  Interventions: Dietary Supplement: Cholecalciferol (Vitamin D3) 70 µg
- placebo (Placebo Comparator)
  Interventions: Other: placebo tablet

INTERVENTIONS:
Dietary Supplement: Cholecalciferol 35 µg per day — Cholecalciferol (Vitamin D3) oral 1 tablet 35 µg per day. Placebo oral 1 tablet per day. In total 35 µg per day.
  In total 2 tablets per day per participant from Baseline to 16 weeks after delivery.
  Arms: Cholecalciferol (Vitamin D3) 35 µg
Other: placebo tablet — placebo 2 tablet, once a day,
  Arms: placebo
Dietary Supplement: Cholecalciferol (Vitamin D3) 70 µg — Cholecalciferol (Vitamin D3) oral 2 tablets each containing 35 µg. In total 70 µg per day.
  In total 2 tablets per day per participant from Baseline to 16 weeks after delivery.
  Arms: Cholecalciferol (Vitamin D3) 70 µg

SUMMARY:
The purpose of this study is to determine whether a daily supplement of vitamin D, taking before and during pregnancy, effects child birth weight, pre- and postpartum complication and bone mineral density during lactation.

ELIGIBILITY:
Inclusion Criteria:

* P-OH25-vitamin D < 50 nmol/l
* Woman age 30-35 years
* In good general health

Exclusion Criteria:

* Infertility
* Intake of 400 IU or more Vitamin D/day
* Cancer
* Alcohol or drug abuse
* Calciummetabolic disturbances
* Spontaneous abortion within last 6 month

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Birth Weight | 0-24 hours after delivery of the child

SECONDARY OUTCOMES:
Post-partum effects of vitamin D supplement on maternal bone mineral density (BMD). | Day 1 to 4 months after delivery.
Infections of the newborn | Day 1 of the child to 16 weeks after birth.
Growth of the newborn measured by weight, crown-heel length and head circumference | Day 1 of the child to 16 weeks after birth
Time to accomplish pregnancy | 0-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Bloch Rasmussen, MD, Principal Investigator — Aarhus University Hospital; Lars Rejnmark, MD, PhD, Drmed., Study Director — Aarhus University Hospital
Locations (1):
- University of Aarhus, Aarhus Universityhospital, Aarhus, Denmark

REFERENCES:
- [Derived] Palacios C, Kostiuk LL, Cuthbert A, Weeks J. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2024 Jul 30;7(7):CD008873. doi: 10.1002/14651858.CD008873.pub5. PMID 39077939